CLINICAL TRIAL: NCT04493437
Title: Future Patient - Telerehabilitation of Atrial Fibrillation Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Collaborators: Aage and Johanne Louis-Hansens Foundation (Unknown); Laboratory of Welfare Technology, Department of Health Science and Technology, AAU (Unknown); Viborg Regional Hospital (Other); Skive Healthcare Center (Unknown); Viborg Healthcare Center (Unknown); University of Aarhus (Other); Department of Photonics Engineering, Technical University of Denmark (Unknown)
Responsible Party: Principal Investigator, Birthe Dinesen, Professor, PhD, Master in Political Science, RN, Head of Laboratory of Welfare Technology - Telehealth & Telerehabilitation, Aalborg University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N-20190059
Record Dates: First submitted 2020-05-28; First posted 2020-07-30 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Telerehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation group A (Experimental): Device: Telerehabilitation Blood pressure (iHealth Neo), weight (iHealth Lina), step counters(Fitbit Inspire & Charge 3), sleep sensor (Emfit QS), tablet (iPad Air 2), and ECG recorder (AliveCor KardiaMobile).
  Interventions: Device: Telerehabilitation
- Telerehabilitation group B (Experimental): Device: Telerehabilitation + rehabilitation at health care center Telerehabilitation: Blood pressure (iHealth Neo), weight (iHealth Lina), step counters(Fitbit Inspire & Charge 3), sleep sensor (Emfit QS), tablet (iPad Air 2), and ECG recorder (AliveCor KardiaMobile).
  Rehabilitation at health care center: The rehabilitation will consist of four closed group sessions focusing on patient education. The groups will consist of both patients and relatives. The program at the health care center will not include any psychological tests or data control. Duration is 4 x 2 hours sessions over a period of 1 month.
  Interventions: Device: Telerehabilitation

INTERVENTIONS:
Device: Telerehabilitation — Blood pressure (iHealth Neo), weight (iHealth Lina), step counters(Fitbit Inspire & Charge 3), sleep sensor (Emfit QS), tablet (iPad Air 2), and ECG recorder (AliveCor KardiaMobile).

SUMMARY:
The idea behind this Future Patient pilot study is to explore and evaluate the feasibility of individualized telerehabilitation technologies and programs for patients with atrial fibrillation (AF).

DETAILED DESCRIPTION:
Objective: To explore the feasibility of individualized telerehabilitation technologies and a program for patients with AF.

Outcome measures:

To evaluate two concepts for telerehabilitation programs and technologies for patients with AF in order to see how these concepts can increase self-management for patients in their rehabilitation process. The following outcome measures are in focus:

Primary outcomes:

* Usability of technologies seen from patients' and healthcare professionals' perspectives
* Test and evaluation of the contents of telerehabilitation programs

Secondary outcomes:

* Measurements of clinical data
* Patients' and relatives' expectations for and experience with participation in the telerehabilitation program
* Healthcare professionals' experience with workflows and collaboration between each other in the telerehabilitation program

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with AF
* Adults ≥ 18 years; no upper age limit
* Patients living in Skive and Viborg Municipality
* Living at home and capable of caring for him/herself
* Basic computer skills or a relative with basic computer skills

Exclusion Criteria:

* Pregnancy
* Lack of ability to cooperate
* Patient does not speak, read and understand Danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2021-05-26 (Actual)

PRIMARY OUTCOMES:
Clinical test of the contents of telerehabilitation programs using interviews | At day 30
  Interviews with patients regarding the use of technology, themes on rehabilitation for AF patients on web portal, and education at healthcare center
Usability test of technologies seen from patients' and healthcare professionals' perspectives | At day 30
  Interviews with patients regarding the user-friendliness of technologies and layout on web portal

SECONDARY OUTCOMES:
Measurements of blood pressure | Every Wednesday: week 1, 2, 3, 4, and 5.
  Evaluation of changes in systolic and diastolic blood pressure measured ones a week
Measurements of pulse | Every Wednesday: week 1, 2, 3, 4, and 5.
  Evaluation of changes in pulse in beats per minut measured ones a week
Measurements of weight | Every Wednesday: week 1, 2, 3, 4, and 5.
  Evaluation of changes in weight in kg measured ones a week
Measurements of electrocardiography (ECG) ECG QT Interval | Every Wednesday: week 1, 2, 3, 4, and 5.
  Evaluation of ECG QT Interval measured ones a week
Measurements of number of steps and sleep | Everyday: week 1, 2, 3, 4, and 5.
  Evaluation of changes in number of steps and sleep measured every day
Interviews on patients' and relatives' expectations for and experience with participation in the telerehabilitation program | At day 30
  Interviews with patients and relatives regarding their experiences with participation in the tele rehabilitation program

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology, Viborg Regional Hospital, Viborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dinesen B, Dam Gade J, Skov Schacksen C, Spindler H, Eie Albertsen A, Dittmann L, Jochumsen M, Svenstrup Moller D. The Danish Future Patient Telerehabilitation Program for Patients With Atrial Fibrillation: Design and Pilot Study in Collaboration With Patients and Their Spouses. JMIR Cardio. 2021 Jul 19;5(2):e27321. doi: 10.2196/27321. PMID 34279239